CLINICAL TRIAL: NCT00443651
Title: An Open-Label, Prospective Study of the Safety of Rituximab in Combination With Other Disease-Modifying Anti-Rheumatic Drugs in Subjects With Active Rheumatoid Arthritis
Brief Title: A Study of the Safety of Rituximab in Combination With Other Anti-Rheumatic Drugs in Subjects With Active Rheumatoid Arthritis
Acronym: SUNDIAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U3924g
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituxan; RA; DMARD; Active Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Anti-Inflammatory Agents

ARMS (2):
- Rituximab 1000 mg (Stage I patients) (Experimental): Stage I patients received 2 doses of rituximab 1000 mg administered intravenously (IV) 14 days apart at the beginning of the study (Days 1 and 15). During Weeks 24 to 40, patients who met disease activity and safety criteria were eligible to receive 2 additional IV infusions of rituximab 1000 mg given 14 days apart. Concomitant non-biological disease-modifying anti-rheumatic drug (DMARD) therapy, at a stable dose and route, was continued during the study, except for protocol defined prohibited DMARDs/combinations.
  Interventions: Drug: Rituximab; Drug: Anti-inflammatory drugs
- Rituximab 500 mg (Stage II patients) (Experimental): Stage II patients received 2 doses of rituximab 500 mg administered intravenously (IV) 14 days apart at the beginning of the study (Days 1 and 15). During Weeks 24 to 40, patients who met disease activity and safety criteria were eligible to receive 2 additional IV infusions of rituximab 500 mg given 14 days apart. Concomitant biological and non-biological disease-modifying anti-rheumatic drug (DMARD) therapy, at a stable dose and route, was continued during the study, except for protocol defined prohibited DMARDs/combinations.
  Interventions: Drug: Rituximab; Drug: Anti-inflammatory drugs

INTERVENTIONS:
Drug: Rituximab — Rituximab was supplied as a concentrate for IV administration at a concentration of 10 mg/mL in 500 mg (50 mL) single-use vials.
Drug: Anti-inflammatory drugs — Each rituximab infusion was preceded by methylprednisolone 100 mg IV. Use of stable doses of oral corticosteroids was permitted (≤ 10 mg of prednisone or equivalent per day) as were stable doses of nonsteroidal anti-inflammatory drugs (NSAIDs).

SUMMARY:
This is a Phase III, open-label study of a total of approximately 560 subjects with active rheumatoid arthritis (RA) who have had an inadequate response to one or more disease-modifying anti-rheumatic drugs (DMARDs). Enrollment in the study was conducted in two stages. In Stage I of the study, approximately 400 subjects receiving non-biological DMARDs (with the exception of methotrexate [MTX] monotherapy or MTX and leflunomide combination therapy) were enrolled. In Stage II of the study, approximately 160 subjects receiving a Federal Drug Administration-approved biological DMARD at the time of screening were enrolled.

ELIGIBILITY:
Inclusion Criteria (Stage I):

* Male or female subjects, between 18 and 80 years of age, who have a documented diagnosis of active rheumatoid arthritis (RA) for ≥ 6 months
* Receiving treatment for RA on an outpatient basis
* Have had an inadequate response to at least one non-biological disease-modifying anti-rheumatic drug (DMARD) and have been receiving this DMARD(s) for ≥ 12 weeks prior to baseline, with stable dose greater than or equal to 4 weeks prior to baseline
* Demonstrated tolerability to currently prescribed DMARDs
* If taking a background corticosteroid, use of the corticosteroid must be at a stable dose during the 4 weeks prior to the first day of treatment with rituximab (Day 1)
* Use of one nonsteroidal anti-inflammatory drug (NSAID) is permitted if the dose is stable for ≥ 2 weeks prior to Day 1

Exclusion Criteria (Stage I):

* Rheumatic autoimmune disease other than RA or significant systemic involvement secondary to RA (including but not limited to vasculitis, pulmonary fibrosis, or Felty's syndrome)
* Functional Class IV as defined by the American College of Rheumatology (ACR) Classification of Functional Status in Rheumatoid Arthritis
* History of or current inflammatory joint disease other than RA or other systemic autoimmune disorder
* Diagnosis of juvenile idiopathic arthritis, or juvenile RA, and/or RA before age 16 years
* Any surgical procedure, including bone/joint surgery/synovectomy (including joint fusion or replacement) within 12 weeks prior to baseline or planned within 24 weeks of enrollment
* Lack of peripheral venous access
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine, or gastrointestinal disorders that, in the investigator's opinion, would preclude subject participation
* Primary or secondary immunodeficiency (history of or currently active), including known history of human immunodeficiency virus (HIV) infection
* Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 4 weeks of baseline or completion of oral antibiotics within 2 weeks prior to baseline
* History of medically significant opportunistic infection
* History of serious recurrent or chronic infection
* History of deep space/tissue infection within 52 weeks prior to baseline
* History of cancer, including solid tumors, hematologic malignancies, and carcinoma in situ (except basal cell and squamous cell carcinoma of the skin that have been excised and cured)
* History of significant cytopenias or other bone marrow disorders
* History of alcohol, drug, or chemical abuse within 24 weeks prior to baseline
* Pregnancy or lactation
* Neuropathies and neurovasculopathies that might interfere with pain evaluation
* Methotrexate (MTX) monotherapy at the time of screening
* Concurrent treatment with MTX and leflunomide in combination
* Concurrent treatment with any biologic agent
* Prior to Day 1, subjects will be discontinued from all DMARDs/combinations that are prohibited in the protocol
* History of a severe allergic or anaphylactic reaction to a biologic agent, or known hypersensitivity to any component of rituximab or to murine proteins
* Previous treatment with an anti-α4 integrin agent
* Previous treatment with any cell-depleting therapies, including investigational agents
* Receipt of any vaccine within 28 days prior to baseline
* Intolerance or contraindications to IV corticosteroids
* Receipt of IV immunoglobulin (IVIG) or Prosorba<TM> column within 6 months prior to baseline
* Any previous treatment with rituximab
* Positive hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody

Inclusion Criteria (Stage II):

* Male or female subjects, between 18 and 80 years of age, who have a documented diagnosis of active RA for ≥ 6 months, diagnosed according to the revised 1987 ACR criteria for the classification of RA
* Receiving treatment for RA on an outpatient basis
* Have had an inadequate response to at least one biologic DMARD and have been receiving this agent at screening and for ≥ 12 weeks prior to baseline, with stable dose greater than or equal to 4 weeks prior to baseline
* Have demonstrated tolerability to currently prescribed DMARDs/biologics
* If taking a background corticosteroid, use of the corticosteroid must be at a stable dose during the 4 weeks prior to baseline
* Use of one NSAID is permitted if the dose is stable for ≥ 2 weeks prior to baseline

Exclusion Criteria (Stage II):

* Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA (including but not limited to vasculitis, pulmonary fibrosis, or Felty's syndrome)
* Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* History of, or current, inflammatory joint disease other than RA or other systemic autoimmune disorder
* Diagnosis of juvenile idiopathic arthritis, or juvenile RA, and/or RA before age 16 years
* Any surgical procedure, including bone/joint surgery/synovectomy (including joint fusion or replacement) within 12 weeks prior to baseline or planned within 24 weeks of randomization
* Lack of peripheral venous access
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine or gastrointestinal disorders that, in the investigator's opinion, would preclude subject participation
* Primary or secondary immunodeficiency (history of or currently active), including known history of HIV infection
* Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of baseline or completion of oral antibiotics within 2 weeks prior to baseline
* History of medically significant opportunistic infection
* History of serious recurrent or chronic infection
* History of deep space/tissue infection within 52 weeks prior to baseline
* History of cancer, including solid tumors, hematologic malignancies, and carcinoma in situ (except basal cell and squamous cell carcinoma of the skin that have been excised and cured)
* History of significant cytopenias or other bone marrow disorders
* History of alcohol, drug, or chemical abuse within 24 weeks prior to baseline
* Pregnancy or lactation
* Neuropathies and neurovasculopathies that might interfere with pain evaluation
* Infliximab monotherapy at the time of screening (infliximab should be in combination with MTX)
* Concurrent treatment with MTX and leflunomide in combination
* Concurrent treatment with more than one biologic agent
* Prior to Day 1, subjects will be discontinued from all DMARDs/combinations that are prohibited in the protocol
* History of a severe allergic or anaphylactic reaction to a biologic agent, or known hypersensitivity to any component of rituximab or to murine proteins
* Previous treatment with an anti-α4 integrin agent
* Previous treatment with any cell-depleting therapies
* Treatment with any investigational agent within 28 days of baseline or 5 half-lives of the investigational drug (whichever is the longer)
* Receipt of any vaccine within 28 days prior to baseline
* Intolerance or contraindications to IV corticosteroids
* Receipt of IVIG or Prosorba<TM> column within 6 months prior to baseline
* Any previous treatment with rituximab
* Positive hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody
* Positive purified protein derivative (PPD) skin test not adequately treated according to Center for Disease Control (CDC) guidelines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micki Klearman, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Rigby WF, Mease PJ, Olech E, Ashby M, Tole S. Safety of rituximab in combination with other biologic disease-modifying antirheumatic drugs in rheumatoid arthritis: an open-label study. J Rheumatol. 2013 May;40(5):599-604. doi: 10.3899/jrheum.120924. Epub 2013 Apr 1. PMID 23547218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 stages. Stage I: Patients with an inadequate response to non-biological disease-modifying antirheumatic drugs (DMARDS) were treated with rituximab 1000 mg. Stage II: Patients with an inadequate response to a biological DMARD were treated with rituximab 500 mg. Both groups continued to receive DMARDs.
Pre-assignment Details: One Stage 1 patient was enrolled but did not receive treatment with rituximab, is not included in the Participant Flow data, and was not included in any of the analyses.
Period: Overall Study
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Started | 401 | 176
Week 24 | 376 | 160
Week 48 | 338 | 134
Completed | 306 (Completed the study or the safety follow-up period.) | 118 (Completed the study or the safety follow-up period.)
Not Completed | 95 | 58
Not completed — Death | 1 | 5
Not completed — Adverse Event | 5 | 6
Not completed — Lost to Follow-up | 18 | 12
Not completed — Patient's/Guardian's Decision | 58 | 30
Not completed — Physician Decision | 13 | 4
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients) | Total
Number analyzed (Participants) | 401 | 176 | 577
Age, Customized [Number; unit: Participants]
  18 - 25 years | 8 | 5 | 13
  26 - 35 years | 22 | 8 | 30
  36 - 45 years | 59 | 26 | 85
  46 - 55 years | 132 | 48 | 180
  56 - 65 years | 133 | 67 | 200
  66 - 75 years | 38 | 19 | 57
  76 - 85 years | 9 | 3 | 12
  > 85 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 154 | 456
  Male | 99 | 22 | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Developing a Serious Adverse Event (SAE) Within 24 Weeks After Receiving the First Course of Rituximab Treatment
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, significantly abnormal laboratory finding, or disease temporally associated with the use of an investigational medical product or other protocol-imposed intervention. An AE was classified as an SAE if it: Resulted in death, persistent or significant disability/incapacity, or congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product; required or prolonged inpatient hospitalization; was life-threatening or considered a significant medical event by the investigator.
Time Frame: From first treatment with rituximab (Day 1) through Week 24
Population: Safety population: All patients who were enrolled in the study and received any study drug (rituximab).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Number analyzed (Participants) | 401 | 176
Percentage of participants | 6.0 | 9.1

2. Secondary Outcome: Percentage of Patients Who Developed a Serious Adverse Event (SAE) During or Within 24 Hours of Rituximab Infusions
Description: The percentage of patients developing a SAE during or within 24 hours of a rituximab infusion is reported separately for each of the 2 infusions in the first course of treatment (Days 1 and 15) and the second course of treatment (optional retreatment during Weeks 24 to 40). See the Primary Outcome Measure for a definition of a SAE.
Time Frame: From start of rituximab treatment through 24 hours
Population: Safety population: All patients who were enrolled in the study and received any study drug (rituximab).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Number analyzed (Participants) | 401 | 176
Percentage of participants
  1st infusion, 1st course of treatment | 0.2 | 0.0
  2nd infusion, 1st course of treatment | 0.0 | 0.0
  1st infusion, 2nd course of treatment | 0.0 | 0.0
  2nd infusion, 2nd course of treatment | 0.0 | 0.0

3. Secondary Outcome: Percentage of Patients Who Developed a Serious Adverse Event (SAE) Within 24 Weeks After Receiving the Second Course (Optional Retreatment) of Rituximab Treatment
Description: as for outcome 1
Time Frame: From start of the second course of rituximab treatment through Week 48
Population: Safety population: All patients who were enrolled in the study and received any study drug (rituximab).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Number analyzed (Participants) | 321 | 147
Percentage of participants | 7.2 | 6.1

4. Secondary Outcome: Percentage of Patients With an Improvement of 20%, 50%, and 70% in American College of Rheumatology (ACR) Scores (ACR20/50/70) From Baseline at Weeks 24 and 48
Description: Improvement must be seen in tender and swollen joint counts and in at least 3 of the following 5 parameters. Patient and physician assessment of patient disease activity (DA) in previous 24 hours on a visual analog scale (VAS, no DA to maximum DA); patient assessment of pain in previous 24 hours on a VAS (none to unbearable); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C reactive protein or, if missing, erythrocyte sedimentation rate.
Time Frame: Baseline to Week 24 and Week 48
Population: Safety population: All patients who were enrolled in the study and received any study drug (rituximab).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Number analyzed (Participants) | 401 | 176
Percentage of participants
  ACR20 at Week 24 | 36.9 | 30.7
  ACR50 at Week 24 | 15.7 | 10.2
  ACR70 at Week 24 | 7.7 | 5.1
  ACR20 at Week 48 | 50.6 | 48.9
  ACR50 at Week 48 | 25.9 | 22.7
  ACR70 at Week 48 | 11.0 | 9.1

5. Secondary Outcome: Percentage of Patients Achieving Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS 28-ESR) Remission and DAS 28-ESR Low Disease Activity Scores at Weeks 24 and 48
Description: DAS 28-ESR was calculated using counts of tender and swollen joints (28 joints, 28TJC and 28SJC), a patient assessment (PA) of disease activity (DA) in previous 24 hours on a visual analog scale (no DA to maximum DA), and ESR at the current visit, using the following formula: 0.56 × 28TJC + 0.28 × 28SJC + 0.70 × ln(ESR) + 0.014 × PADA. The DAS 28-ESR score ranges from 0 to 10, with higher scores indicating more rheumatoid arthritis. DAS28-ESR Remission was defined as a DAS 28-ESR score of < 2.6. DAS28-ESR Low Disease Activity was defined as a DAS28-ESR score of ≤ 3.2.
Time Frame: Week 24 and Week 48
Population: Safety population: All patients who were enrolled in the study and received any study drug (rituximab). There were 401 patients in the rituximab 1000 mg and 176 patients in the 500 mg safety populations. n = number of patients with non-missing DAS28-ESR last observation carried forward scores at Weeks 24 and 48 in the safety populations.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Number analyzed (Participants) | 401 | 176
Percentage of participants
  DAS 28-ESR Remission at Week 24 (n=391, 171) | 8.4 | 6.4
  DAS 28-ESR Low DA at Week 24 (n=391, 171) | 15.6 | 11.7
  DAS 28-ESR Remission at Week 48 (n=389, 172) | 12.6 | 7.0
  DAS 28-ESR Low DA at Week 48 (n=389, 172) | 23.4 | 22.1

6. Secondary Outcome: Percentage of Patients With European League Against Rheumatism (EULAR) Good and Moderate Responses at Weeks 24 and 48
Description: Improvement in the post-baseline DAS 28-ESR score from baseline was used to determine the EULAR responses of moderate response and good response. The DAS 28-ESR score ranges from 0 to 10, with higher scores indicating more rheumatoid arthritis. For a post-baseline score ≤ 3.2, an improvement > 0.6 to ≤ 1.2 was a moderate response and ≥ 1.2 a good response. For a post-baseline score > 3.2 to ≤ 5.1, an improvement > 0.6 was a moderate response. For a post-baseline score > 5.1, an improvement ≥ 1.2 was a moderate response. A good response could not be achieved for post-baseline scores > 3.2.
Time Frame: Baseline to Week 24 and Week 48
Population: Safety population: All patients who were enrolled in the study and received any study drug (rituximab).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Number analyzed (Participants) | 401 | 176
Percentage of participants
  Good EULAR Response at Week 24 | 13.7 | 9.1
  Moderate EULAR Response at Week 24 | 39.2 | 34.1
  Good EULAR Response at Week 48 | 21.2 | 18.2
  Moderate EULAR Response at Week 48 | 44.1 | 43.8

7. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Change From Baseline at Weeks 24 and 48
Description: The HAQ-DI assesses how well the patient is able to perform 8 activities: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. The patient answers 20 questions with 1 of 4 responses with the past week as the time frame: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The highest score for any question in a category determines the category score. The total score ranges from 0 (no disability) to 3 (completely disabled). A negative change score indicates improvement.
Time Frame: Baseline to Week 24 and Week 48
Population: Safety population: All patients who were enrolled in the study and received any study drug (rituximab).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Number analyzed (Participants) | 389 | 172
Units on a scale
  Week 24 | -0.28 (0.474) | -0.28 (0.495)
  Week 48 | -0.33 (0.508) | -0.32 (0.512)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were recorded from the time when informed consent was obtained until Week 48, Week 4 of the safety follow-up (SFU) period, or early discontinuation. Beyond Week 4 of the SFU period, only serious or infectious AEs were recorded.
Description: Safety population: All patients who were enrolled in the study and received any study drug (rituximab).
Arm/Group | Rituximab 1000 mg (Stage I Patients) | Rituximab 500 mg (Stage II Patients)
Serious Adverse Events (participants affected / at risk) | 48/401 | 27/176
Other Adverse Events (participants affected / at risk) | 278/401 | 128/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (Stage I Patients) (N=401) | Rituximab 500 mg (Stage II Patients) (N=176)
Chest pain (General disorders) | 4 | 1
Pelvic mass (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 4 | 1
Bronchitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Colitis ischemic (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Gastritis hemorrhagic (Gastrointestinal disorders) | 0 | 1
Yolk sac tumor site unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Hemicephalalgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Microcytic anemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (Stage I Patients) (N=401) | Rituximab 500 mg (Stage II Patients) (N=176)
Nausea (Gastrointestinal disorders) | 31 | 22
Vomiting (Gastrointestinal disorders) | 21 | 8
Diarrhoea (Gastrointestinal disorders) | 25 | 10
Oedema peripheral (General disorders) | 13 | 10
Upper respiratory tract infection (Infections and infestations) | 51 | 27
Sinusitis (Infections and infestations) | 45 | 23
Urinary tract infection (Infections and infestations) | 45 | 15
Bronchitis (Infections and infestations) | 35 | 12
Influenza (Infections and infestations) | 13 | 9
Contusion (Injury, poisoning and procedural complications) | 5 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 50 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 12
Headache (Nervous system disorders) | 38 | 25
Depression (Psychiatric disorders) | 20 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 10
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Rash (Skin and subcutaneous tissue disorders) | 28 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 11
Hypertension (Vascular disorders) | 28 | 14
Flushing (Vascular disorders) | 18 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.